CLINICAL TRIAL: NCT02952963
Title: Effect of Bile Acids and Bile Acid Sequstrants on GLP-1 Secretion After Roux-en-Y Gastric Bypass
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Maria Saur Svane, MD, Principal Investigator, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IJ-GALDE3-16
Record Dates: First submitted 2016-11-01; First posted 2016-11-02 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Severe Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Chenodeoxycholic Acid; Colesevelam Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chenodeoxycholic Acid (Experimental): Chenodeoxycholic Acid (1250 mg) dissolved in 200 ml water. Here after 50 ml clean water.
  Interventions: Drug: Chenodeoxycholic Acid
- Chenodeoxycholic Acid and Colesevelam (Experimental): Chenodeoxycholic Acid (1250 mg) and Colesevelam (3,75 g) dissolved in 200 ml water. Here after 50 ml clean water.
  Interventions: Drug: Chenodeoxycholic Acid; Drug: Colesevelam

INTERVENTIONS:
Drug: Chenodeoxycholic Acid
Drug: Colesevelam
  Arms: Chenodeoxycholic Acid and Colesevelam

SUMMARY:
The purpose of this study is to examine the efffects of bile acid and bile acids sequestrants on GLP-1 secretion, in patients after Roux-en-Y gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated RYGB performed minimum 3 months prior to the study.
* Fasting glucose < 7,0 mM, HbA1c < 48 mmol/mol 3 months after RYGB

Exclusion Criteria:

* Fasting plasma glucose > 7,0 mM, HbA1c > 48 mmol/mol 3 months after RYGB
* Dysregulated thyroid diseases, use of antithyroid treatment.
* Late diabetic complications as retinopathy, renal insufficiency, neuropathy or previous pancreatitis.
* Complications to RYGB. Documented reactive hypoglycaemia, severe dumping (vomiting, diarrhea, severe abdominal pain after food intake)
* Cholecystectomy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-10; Primary Completion 2017-12 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
GLP-1 secretion (evaluated by iAUC) | -10, 0, 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180 and 240 minutes after medicin intake.

SECONDARY OUTCOMES:
Glucose levels | -10, -5, 0, 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180 and 240 minutes
PYY secretion | -10, 0, 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180 and 240 minutes
Glucagon secretion | -10, 0, 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180 and 240 minutes
GIP secretion | -10, 0, 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180 and 240 minutes
Insulin secretion | -10, -5, 0, 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180 and 240 minutes
C-peptide secretion | -10, -5, 0, 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180 and 240 minutes
CCK secretion | -10, 0, 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180 and 240 minutes
Total ghrelin | -10, 0, 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180 and 240 minutes
Total bile acid secretion | -10, 0, 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180 and 240 minutes
Bile acids fractions / FGF-19 concentrations | -10, 0, 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180 and 240 minutes
Appetite measurements (VAS-score) | -10, 30, 60, 120, 180 and 240 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, DK, Denmark

IPD SHARING:
Plan to Share IPD: Yes